CLINICAL TRIAL: NCT03660059
Title: A Randomized, Double-Blind, Placebo-Controlled Confirmatory Study of the Safety and Efficacy of ASP015K in Patients With Rheumatoid Arthritis (RA) Who Had an Inadequate Response or Intolerance to MTX
Brief Title: A Study to Assess Safety and Efficacy of ASP015K in Participants With Rheumatoid Arthritis (RA) Who Had an Inadequate Response or Intolerance to Methotrexate (MTX)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 015K-CL-CNA3; CTR20181199 (Registry Identifier: ChinaDrugTrials.org.cn)
Record Dates: First submitted 2018-08-26; First posted 2018-09-06 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: rheumatoid arthritis (RA); efficacy; ASP015K; Peficitinib; safety
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — peficitinib; Antirheumatic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASP015K 100 mg (Experimental): Participants will receive 100 milligrams (mg) of ASP015K once daily after breakfast for 52 weeks.
  Interventions: Drug: Peficitinib; Drug: Disease-modifying antirheumatic drugs (DMARDs)
- ASP015K 150 mg (Experimental): Participants will receive 150 mg of ASP015K once daily after breakfast for 52 weeks.
  Interventions: Drug: Peficitinib; Drug: Disease-modifying antirheumatic drugs (DMARDs)
- Placebo/ASP015K (Placebo Comparator): Participants will receive placebo for 24 weeks, then either 100 mg or 150 mg of ASP015K for 28 weeks as determined randomly at Week 0 in advance.
  Interventions: Drug: Peficitinib; Drug: Plaebo; Drug: Disease-modifying antirheumatic drugs (DMARDs)

INTERVENTIONS:
Drug: Peficitinib — Oral
  Other Names: ASP015K
Drug: Plaebo — Oral
  Arms: Placebo/ASP015K
Drug: Disease-modifying antirheumatic drugs (DMARDs) — As necessary concomitant medications, DMARDs listed below will be administered orally unless specified.
  For subjects who are inadequate responders to methotrexate (MTX): MTX. For subjects who are intolerant of MTX: either of DMARDs listed; hydroxychloroquine, salazosulfapyridine, gold (injection or oral), D-penicillamine, lobenzarit, actarit, bucillamine and iguratimod.

SUMMARY:
The purpose of this study is to verify the superiority of ASP015K in combination with MTX or with other disease-modifying antirheumatic drugs (DMARDs) over placebo in terms of efficacy in participants with rheumatoid arthritis (RA) who had an inadequate response or intolerance to MTX, as measured by the American College of Rheumatology (ACR) 20 response rate at Week 24.

This study will also evaluate the pharmacokinetics and safety of ASP015K as well as efficacy and safety of long-term treatment with ASP015K (52 weeks).

DETAILED DESCRIPTION:
Participants will be randomized in a 1:1:1 ratio to the ASP015K dose-A group, ASP015K dose-B group or placebo group at Week 0.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a man or woman and considered to be an adult, according to the local legal definition, at the time of informed consent.
* Subject has RA diagnosed according to the 1987 American College of Rheumatology (ACR) criteria or the 2010 American College of Rheumatology/European League against Rheumatism (ACR/EULAR) criteria.
* Subject did not receive the following drugs, or received the drugs with stable dosage for at least 28 days prior to the baseline (start of treatment) for RA treatment: Non-steroidal anti-inflammatory drugs (NSAIDs; excluding topical formulations), oral morphine or equivalent opioid analgesics (≤ 30 mg/day), acetaminophen, or oral corticosteroids (≤ 10 mg/day in prednisolone equivalent).
* Subject has active RA as evidenced by both of the following:

  * ≥ 6 tender/painful joints (using 68-joint assessment)
  * ≥ 6 swollen joints (using 66-joint assessment)
* Subject has CRP > 0.50 mg/dL. The re-test of CRP will be allowed, if the subject's CRP value at the time of screening test is more than 0.30 mg/dL and also his/her most recent CRP value which was carried out up to 90 days before the date of screening test was more than 0.5 mg/dL.
* Subject meets the ACR 1991 Revised Criteria for the Classification of Global Functional Status in RA Class I, II, or III.
* Subject has inadequate response or intolerance for MTX.
* For inadequate responder to MTX, subject has had regular use of MTX for at least 90 days prior to screening at a dose that, in accordance with local clinical practice, is considered acceptable to adequately assess clinical response. The dose of MTX must have been a stable, unchanging oral dose of 7.5 to 20 mg/week (or the equivalent injectable dose) for at least the 28 days prior to screening. Subject is able to continue stable dose of MTX from at least 28 days prior to screening until the end of the administration period of study drug.
* For subject who is intolerant of MTX, subject has had regular use of the following DMARDs, and when the following DMARDs are concomitantly administered to subject, the drugs must be administered for at least 90 days prior to screening, and must be stable from at least 28 days prior to screening until the end of the administration period of study drug.

  * Hydroxychloroquine
  * Salazosulfapyridine
  * Gold
  * D-penicillamine
  * Lobenzarit
  * Actarit
  * Bucillamine
  * Iguratimod

Exclusion Criteria:

* Subject has received a biologic DMARD within the specified period:

  * Anakinra: within 28 days prior to baseline
  * Etanercept: within 28 days prior to baseline
  * Adalimumab, infliximab: within 56 days prior to baseline
  * Golimumab, certolizumab pegol: within 70 days prior to baseline
  * Abatacept, tocilizumab: within 84 days prior to baseline
  * Denosumab: within 150 days prior to baseline
  * Rituximab: within 180 days prior to baseline
* Subject has inadequate response to at least 3 biologic DMARDs.
* Subject has received a non-biologic DMARD listed below or other drugs used in the treatment of RA within 28 days prior to baseline. Leflunomide is prohibited within 90 days prior to baseline. Alternatively, leflunomide is prohibited at least 28 days prior to baseline if washout with cholestyramine for at least 17 days is completed within 28 days prior to baseline. However, topical drugs other than those for the treatment of RA may be used concomitantly.

  * Leflunomide
  * Tacrolimus
  * Cyclosporine
  * Cyclophosphamide
  * Azathioprine
  * Minocycline
  * Mizoribine
* Subject has received Chinese herbal medicines listed below or other herbal drugs used in the treatment of RA within 28 days prior to baseline.

  * Tripterygium wilfordii
  * Total glucosides of paeony
  * Tsuduranine
* Subject has received tofacitinib, baricitinib or other JAK inhibitor (including other investigational drugs).
* Subject has received intra-articular, intravenous, intramuscular, or endorectal (including suppositories for anal diseases) corticosteroid within 28 days prior to baseline.
* Subject has participated in any study of ASP015K and has received ASP015K or placebo.
* Subject has received other investigational drugs within 90 days or within 5 half-lives, whichever is longer, prior to baseline.
* Subject has received plasma exchange therapy within 60 days prior to baseline.
* Subject has undergone joint drainage, has received local anesthesia and nerve block, or has received articular cartilage protectant (such as glucosamine sulfate, chondroitin sulfate these DMORD medicine) at the assessed joint within 28 days prior to baseline.
* Subject has undergone surgery and has residual effects in the assessed joints or is scheduled to undergo surgery that may affect the study evaluation of the assessed joints.
* Subject is diagnosed as inflammatory arthritis (psoriatic arthritis, ankylosing spondylitis, SLE, sarcoidosis, etc.) other than RA.
* Subject has any of the following laboratory values:

  * Hemoglobin < 9.0 g/dL
  * Absolute neutrophil count < 1000/μL
  * Absolute lymphocyte count < 800/μL
  * Platelet count < 75000/μL
  * Alanine aminotransferase (ALT) ≥ 2 × upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) ≥ 2 × ULN
  * Total bilirubin (TBL) ≥ 1.5 × ULN
  * Estimated glomerular filtration rate (eGFR) ≤ 40 mL/min as measured by the MDRD method
  * β-D-glucan > ULN
* Subject has a history of or concurrent active tuberculosis (TB). Eligibility criteria for TB are tabulated below:
* Subject meets any of the following in terms of infection except for TB:

  * History of or concurrent severe herpes zoster (associated with Hunt syndrome or having ulcerative lesions) or disseminated herpes zoster
  * History of multiple recurrences (at least twice) of localized herpes zoster
  * Serious infection requiring hospitalization within 90 days prior to baseline
  * Subject has received intravenous antibiotics within 90 days prior to baseline. (However, prophylactic antibiotics are allowed.)
  * Subject with high risk of infection (e.g., subject with urinary catheter)
* Subject has a history of or concurrent interstitial pneumonia and inappropriate to participate in this study.
* Subject has a history of or concurrent malignant tumor (except for successfully treated basal cell carcinoma).
* Subject has received live or live attenuated virus vaccination within 56 days prior to baseline. (Inactivated vaccines including influenza and pneumococcal vaccines are allowed.)
* Subject has any ongoing severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, neurological, infectious, or autoimmune disease except for RA (excluding Sjogren's syndrome and chronic thyroiditis), or any ongoing illness which would make the subject unsuitable for the study.
* Subject has a history of clinically significant allergy. (Clinically significant allergy includes allergies such as systemic urticaria induced by specific antigens and drugs, anaphylaxis, and allergy associated with shock necessitating hospitalized treatment.)
* Subject has received medications that are CYP3A substrates with narrow therapeutic range within 14 days prior to baseline. These medications include: dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, temsirolimus, and disopyramide.
* Subject has concurrent cardiac failure, defined as New York Heart Association (NYHA) classification Class III or higher, or a history of it.
* Subject has concurrent prolonged QT syndrome or a history of it. Subject has prolonged QT interval (defined as QTc ≥ 500 msec. Subject has QTc ≥ 500 msec at retest will be excluded).
* Subject has congenital short QT syndrome or a history of it. Subject has shortened QT interval (defined as QTc < 330 msec. Subject has QTc < 330 msec at retest will be excluded).
* Subject has a history of positive HIV infection.
* Female subject is pregnant or might be pregnant, is nursing, wishes to conceive for a period running from the time informed consent is given within 60 days after end of treatment, or for whom the possibility of pregnancy cannot be ruled out as a result of the serum pregnancy test given at the time of screening.
* Male subject cannot practice at least 2 types of contraception from the time of informed consent to 90 days after end of treatment, or subject is a woman with childbearing potential who cannot practice at least 2 types of contraception from the time of informed consent to 60 days after end of treatment.
* Male subject does not agree not to donate sperm starting at informed consent and through the treatment period and for at least 90 days after final study drug administration. Female subject who do not agree not to donate ova starting at informed consent through the treatment period and for 60 days after final study drug administration.
* Subject has a history or complication of lymphatic diseases such as lymphoproliferative disorder, lymphoma, and leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology (ACR)20 response rate at Week 24 | At Week 24
  The ACR20 response requires that all criteria from (1) to (3) be met compared with Week 0 (baseline); (1), Tender Joint Count (TJC) >= 20% reduction; (2), Swollen Joint Count (SJC) >= 20% reduction;(3) >= 20% improvement in three or more of the following five parameters - [1] subject's assessment of pain, [2] Subject's Global Assessment of Arthritis (SGA), [3] Physician's Global Assessment of Arthritis (PGA), [4] health assessment questionnaire-disability index (HAQ-DI), [5] acute phase reactant (C-reactive protein (CRP) or erythrocyte sedimentation rate (ESR)).

SECONDARY OUTCOMES:
ACR20 response rate | Up to Week 52
  The ACR20 response requires that all criteria from (1) to (3) be met compared with Week 0 (baseline); (1), Tender Joint Count (TJC) >= 20% reduction; (2), Swollen Joint Count (SJC) >= 20% reduction;(3) >= 20% improvement in three or more of the following five parameters - [1] subject's assessment of pain, [2] Subject's Global Assessment of Arthritis (SGA), [3] Physician's Global Assessment of Arthritis (PGA), [4] health assessment questionnaire-disability index (HAQ-DI), [5] acute phase reactant (C-reactive protein (CRP) or erythrocyte sedimentation rate (ESR)).
ACR50 response rate | Up to Week 52
  The ACR50 response indicates a 50% improvement in all criteria used in the ACR20 assessment.
ACR70 response rate | Up to Week 52
  The ACR70 response indicates a 70% improvement in all criteria used in the ACR70 assessment.
Change from baseline in disease activity score (DAS) 28-C-reactive protein (CRP) scores | From baseline (Week 0) to Week 52
  DAS28-CRP will be calculated using data from TJC (28 joints), SJC (28 joints), CRP and SGA with the formula; DAS28-CRP = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP + 1) + 0.014 x SGA + 0.96
Change from baseline in DAS28- erythrocyte sedimentation rate (ESR) scores | From baseline (Week 0) to Week 52
  DAS28-ESR will be calculated using data from TJC (28 joints), SJC (28 joints), ESR and SGA with the formula; DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 x SGA
Change from baseline in Tender Joint Count (TJC) (68 joints) | From baseline (Week 0) to Week 52
  The investigator/sub-investigator will examine the participant for tender joints, assessing the 68 joints and confirm the location of each tender joint.
Change from baseline in Swollen Joint Count (SJC) (66 joints) | From baseline (Week 0) to Week 52
  The investigator/sub-investigator will examine the participants for swollen joints, assessing the 66 joints, where hip joints are excluded from 68 joints, and confirm the location of the swollen joints.
Percentage of participants achieving DAS28-CRP scores for remission | Up to Week 52
  Percentage of participants with DAS28 scores less than 2.6.
Percentage of participants achieving DAS28-ESR scores for remission | Up to Week 52
  Percentage of participants with DAS28 scores less than 2.6.
Percentage of participants achieving low disease activity by DAS28-CRP | Up to Week 52
  DAS28 score exceeding 5.1 is considered high disease activity; 3.2 to 5.1, moderate disease activity; less than 3.2, low disease activity.
Percentage of participants achieving low disease activity by DAS28-ESR | Up to Week 52
  DAS28 score exceeding 5.1 is considered high disease activity; 3.2 to 5.1, moderate disease activity; less than 3.2, low disease activity.
Change from baseline in CRP | From baseline (Week 0) to Week 52
  CRP will be measured with blood samples.
Change from baseline in ESR | From baseline (Week 0) to Week 52
  ESR will be measured with blood samples.
Percentage of participants with good European League Against Rheumatism (EULAR) response | Up to Week 52
  Based on DAS28 scores and changes in DAS28 scores before and after treatment with the study drug, EULAR Response Criteria categorize response to treatment as "No response", "Moderate response," or "Good response."
Percentage of participants with good or moderate EULAR response | At Week 52
  Based on DAS28 scores and changes in DAS28 scores before and after treatment with the study drug, EULAR Response Criteria categorize response to treatment as "No response", "Moderate response," or "Good response."
Percentage of participants achieving ACR/EULAR remission | At Week 52
  If all of the following 4 parameters are fulfilled, it is defined as remission: TJC ≤ 1, SJC ≤ 1, CRP ≤ 1 mg/dL, SGA ≤ 1 cm (on a visual analog scale (VAS) of 0 - 100 mm).
Percentage of participants achieving Simplified Disease Activity Index (SDAI) remission (SDAI score ≤ 3.3) | Up to Week 52
  SDAI score will be calculated with formula SDAI = TJC + SJC + SGA + PGA + CRP. SDAI score exceeding 26 is considered high disease activity; exceeding 11 and not greater than 26, moderate disease activity; exceeding 3.3 and not greater than 11, low disease activity.
Change from baseline in SDAI score | From baseline (Week 0) to Week 52
  Change from baseline (Week 0) in SDAI score will be calculated.
Change from baseline in Physician's Global Assessment of Arthritis (PGA) (VAS) | From baseline (Week 0) to Week 52
  The investigator/sub-investigator assesses the participant's disease activity on a VAS of 0 - 100 mm on the physician assessment table.
Change from baseline in SGA (VAS) | From baseline (Week 0) to Week 52
  The participant assesses his/her own disease activity on a VAS of 0 - 100 mm on the questionnaire form.
Change from baseline in participant's assessment of pain (VAS) | From baseline (Week 0) to Week 52
  The participant assesses his/her own pain severity on a VAS of 0 - 100 mm on the questionnaire form.
Incidence of participant withdrawal due to the lack of efficacy | Up to Week 56
  Number of participants who withdraw from this study due to the lack of efficacy.
Change from baseline in health assessment questionnaire-disability index (HAQ-DI) score | From baseline (Week 0) to Week 52
  The HAQ-DI measure shave eight dimensions of functional activity: pruning, dressing, rising, eating, walking, personal hygiene, reach, grip, and other routine activities. Each item has 4 degrees ranging from 0 to 3. "0" refers to "no functional difficulty", "1" to a bit of functional difficulty, "2" to very much functional difficulty, and "3" to no ability to work. HAQ-DI score 0-1 means mild to moderate functional difficulty; 1-2 means moderate to severe disability; and 2-3 means generally severe disability.
Change from baseline in Short Form Health Survey - 36 questions, version 2 (SF-36v2)® score | From baseline (Week 0) to Week 52
  SF-36v2 is a validated instrument used to measure general physical and mental health status via assessment of 8 domains - physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental. The SF-36 is scored using norm-based scoring procedures and scores ranging from 0-100; higher scores represent better health-related quality of life.
Change from baseline in Work Productivity and Activity Impairment Questionnaire (WPAI) score | From baseline (Week 0) to Week 52
  WPAI produces four types of scores: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment. The WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Pharmacokinetics (PK) of ASP015K in plasma: post-dose concentration | 2 hours post-dose at either Week 4 or Week 8
  Post-dose concentration will be derived from the PK plasma samples collected.
PK of ASP015K in plasma: trough concentration (Ctrough) | Up to Week 52
  Ctrough will be derived from the PK plasma samples collected.
Safety assessed by incidence of adverse events (AEs) | Up to Week 56
  An AE is defined as any untoward medical occurrence after the signing of informed consent form in a participant administered a study drug or who has undergone study procedures and which does not necessarily have a causal relationship with this treatment.
Number of participants with vital sign abnormalities and/or AEs | Up to Week 56
  Number of participants with potentially clinically significant vital sign values.
Number of participants with body weight abnormalities and/or AEs | Up to Week 56
  Number of participants with potentially clinically significant body weight values.
Number of participants with 12-lead electrocardiogram (ECG) abnormalities and/or AEs | Up to Week 52
  Number of participants with potentially clinically significant 12-ECG values.
Number of participants with central ECG abnormalities and/or AEs | Up to Week 8
  Number of participants with potentially clinically significant central ECG observations. Central ECG will be measured before and 2 hours after study drug administration.
Number of participants with chest radiography abnormalities and/or AEs | Up to Week 52
  Number of participants with potentially clinically significant chest radiography observations.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Inc
Locations (43):
- China (33):
  - Site CN00048, Anhui
  - Site CN00045, Beijing
  - Site CN00054, Beijing
  - Site CN00050, Bengbu
  - Site CN00061, Changchun
  - Site CN00032, Changsha
  - Site CN00076, Chenzhou
  - Site CN00071, Guangdong
  - Site CN00016, Guangzhou
  - Site CN00052, Guangzhou
  - Site CN00063, Guangzhou
  - Site CN00072, Guangzhou
  - Site CN00058, Inner Mongolia
  - Site CN00074, Jieyang
  - Site CN00028, Jilin
  - Site CN00069, Jining
  - Site CN00064, Jiujiang
  - Site CN00046, Kunming
  - Site CN00060, Nanjing
  - Site CN00070, Nanjing
  - Site CN00068, Ningbo
  - Site CN00075, Pingxiang
  - Site CN00066, Qingdao
  - Site CN00056, Shanghai
  - Site CN00047, Shantou
  - Site CN00053, Sichuan
  - Site CN00057, Tianjin
  - Site CN00062, Tianjin
  - Site CN00059, Wuhan
  - Site CN00067, Xining
  - Site CN00065, Xuzhou
  - Site CN00073, Zhengzhou
  - Site CN00049, Zhuzhou
- South Korea (5):
  - Site KR00037, Gwangju
  - Site KR00036, Incheon
  - Site KR00033, Seoul
  - Site KR00034, Seoul
  - Site KR00035, Seoul
- Taiwan (5):
  - Site TW00022, Taichung
  - Site TW00023, Taichung
  - Site TW00024, Taichung
  - Site TW00025, Taipei
  - Site TW00026, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Yang Y, Li J, Liu J, Liu L, Wang Y, Hu J, Li Z, Gu J, Zhang X, Xiao Z, Zheng J, Liu L, Li Z, Wei JC. Safety and efficacy of peficitinib in Asian patients with rheumatoid arthritis who had an inadequate response or intolerance to methotrexate: results of a multicenter, randomized, double-blind, placebo-controlled phase 3 study. Lancet Reg Health West Pac. 2023 Oct 18;42:100925. doi: 10.1016/j.lanwpc.2023.100925. eCollection 2024 Jan. PMID 38357391
- See also: Link to results on the Astellas Clinical Study Results website — https://www.clinicaltrials.astellas.com/study/015K-CL-CNA3/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14521&tenant=MT_AST_9011